CLINICAL TRIAL: NCT00014508
Title: A Phase II Trial Of Autologous Stem Cell Transplant Followed By Mini-Allogeneic Stem Cell Transplant In Lieu Of Standard Allogeneic Bone Marrow Transplantation For Treatment Of Multiple Myeloma
Brief Title: Chemotherapy and Peripheral Stem Cell Transplantation in Treating Patients With Multiple Myeloma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000068551; ECOG-E4A98
Record Dates: First submitted 2001-04-10; First posted 2003-01-27 (Estimated); Last update posted 2023-06-22 (Actual); Status verified 2023-06

CONDITIONS: Multiple Myeloma and Plasma Cell Neoplasm
Keywords: refractory multiple myeloma; stage I multiple myeloma; stage II multiple myeloma; stage III multiple myeloma
MeSH Terms: conditions — Multiple Myeloma; Neoplasms, Plasma Cell | interventions — sargramostim; Cyclophosphamide; Cyclosporine; fludarabine phosphate; Melphalan; Peripheral Blood Stem Cell Transplantation

INTERVENTIONS:
Biological: sargramostim
Drug: cyclophosphamide
Drug: cyclosporine
Drug: fludarabine phosphate
Drug: melphalan
Procedure: peripheral blood stem cell transplantation

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop cancer cells from dividing so they stop growing or die. Peripheral stem cell transplantation may be able to replace immune cells that were destroyed by chemotherapy. Sometimes the transplanted cells are rejected by the body's tissues. Peripheral stem cell transplantation with the person's own stem cells followed by donor peripheral stem cell transplantation may prevent this from happening.

PURPOSE: Phase II trial to study the effectiveness of combining chemotherapy with autologous peripheral stem cell transplantation and donor peripheral stem cell transplantation in treating patients who have multiple myeloma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the incidence of early mortality in patients with multiple myeloma treated with melphalan and autologous peripheral blood stem cell (PBSC) transplantation followed by fludarabine, cyclophosphamide, and allogeneic PBSC transplantation.
* Determine the incidence of early allogeneic graft failure (before day 100 after allogeneic PBSC transplantation) and the incidence of severe acute graft-versus-host disease (GVHD) in patients treated with this regimen.
* Determine the toxicity of this regimen in these patients.
* Determine the overall and disease-free survival of patients treated with this regimen.
* Correlate changes in the T-cell population with clinical outcome, such as survival, in patients treated with this regimen.
* Correlate changes in the T-cell population with the incidence of GVHD, use of immunosuppressive agents, and effects of fludarabine in patients treated with this regimen.
* Determine the degree of chimerism after allogeneic PBSC transplantation and the time course over which it is established in patients treated with this regimen.

OUTLINE: This is a multicenter study.

Patients receive melphalan IV over 15 minutes on day -1. Autologous peripheral blood stem cells (PBSCs) are reinfused on day 0. Patients also receive sargramostim (GM-CSF) subcutaneously (SC) or IV over at least 30 minutes daily beginning on day 1 and continuing until blood counts recover. Beginning 100-182 days after autologous PBSC transplantation, patients receive fludarabine IV over 30 minutes on days -6 to -2 and cyclophosphamide IV over 1-2 hours on days -3 and -2. Allogeneic PBSCs are infused on day 0. Patients may receive a second allogeneic PBSC infusion on day 1. Patients also receive GM-CSF SC or IV over at least 30 minutes daily beginning on day 1 and continuing until blood counts recover. Cyclosporine is administered IV or orally twice daily as graft-versus-host disease (GVHD) prophylaxis, beginning on day -1 and continuing until day 60, followed by a taper in the absence of GVHD.

Patients are followed for 5 years.

PROJECTED ACCRUAL: A total 19-46 patients will be accrued for this study within 3 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of multiple myeloma meeting 1 of the following criteria:

  * Bone marrow plasmacytosis with at least 10% plasma cells
  * Sheets of plasma cells
  * Biopsy-proven plasmacytoma
* Meets at least 1 of the following criteria:

  * Presence of myeloma (M)-protein in the serum
  * Presence of M-protein in the urine
  * Radiographic evidence of osteolytic lesions

    * Generalized osteoporosis allowed if at least 20% plasma cells in bone marrow
* No non-secretory myeloma

  * Prior M-protein in serum or urine allowed provided patient is now in complete remission
* Must be receiving conventional-dose chemotherapy as initial therapy or as salvage therapy
* Must have HLA-A, -B, and -DR genotypically identical sibling donor

PATIENT CHARACTERISTICS:

Age:

* 18 to 70

Performance status:

* ECOG 0-2

Life expectancy:

* Not specified

Hematopoietic:

* See Disease Characteristics

Hepatic:

* AST no greater than 3 times upper limit of normal
* Bilirubin less than 2.0 mg/dL

Renal:

* Not specified

Cardiovascular:

* LVEF greater than 40% at rest if symptomatic cardiac disease is present

Pulmonary:

* DLCO greater than 50% of predicted (corrected for hemoglobin) if symptomatic pulmonary disease is present

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* No prior autologous or allogeneic peripheral blood stem cell or bone marrow transplantation

Chemotherapy:

* See Disease Characteristics
* More than 28 days since prior chemotherapy (including primary chemotherapy for hematopoietic stem cell collection)
* No other concurrent cytotoxic chemotherapy between autologous and allogeneic transplantation

Endocrine therapy:

* Prior dexamethasone or other corticosteroids allowed
* Concurrent corticosteroids between autologous and allogeneic transplantation allowed

Radiotherapy:

* Concurrent radiotherapy between autologous and allogeneic transplantation allowed

Surgery:

* Not specified

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2001-11-19 (Actual); Primary Completion 2007-02 (Actual); Study Completion 2011-05-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Neal Flomenberg, MD, Study Chair — Sidney Kimmel Cancer Center at Thomas Jefferson University
Locations (12):
- United States (12):
  - Baptist Cancer Institute - Jacksonville, Jacksonville, Florida
  - Mayo Clinic - Jacksonville, Jacksonville, Florida
  - Cancer Center at Tufts - New England Medical Center, Boston, Massachusetts
  - Beth Israel Deaconess Medical Center, Boston, Massachusetts
  - Mayo Clinic Cancer Center, Rochester, Minnesota
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey at UMDNJ - Robert Wood Johnson Medical School, New Brunswick, New Jersey
  - MBCCOP-Our Lady of Mercy Cancer Center, The Bronx, New York
  - Ireland Cancer Center at University Hospitals of Cleveland and Case Western Reserve University, Cleveland, Ohio
  - MetroHealth's Cancer Care Center at MetroHealth Medical Center, Cleveland, Ohio
  - Penn State Cancer Institute at Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - Abramson Cancer Center at the University of Pennsylvania, Philadelphia, Pennsylvania

REFERENCES:
- [Background] Vesole DH, Zhang L, Flomenberg N, Greipp PR, Lazarus HM, Huff CA; ECOG Myeloma and BMT Committees. A Phase II trial of autologous stem cell transplantation followed by mini-allogeneic stem cell transplantation for the treatment of multiple myeloma: an analysis of Eastern Cooperative Oncology Group ECOG E4A98 and E1A97. Biol Blood Marrow Transplant. 2009 Jan;15(1):83-91. doi: 10.1016/j.bbmt.2008.10.030. PMID 19135946